CLINICAL TRIAL: NCT00678171
Title: A Pilot Study to Evaluate an OP-1 Putty Spinal System and an Autograft Spinal System in Patients Requiring Transforaminal Lumbar Interbody Fusion of the Spine
Brief Title: A Pilot Study to Evaluate an Osteogenic Protein 1 (OP-1) Putty Spinal System and an Autograft Spinal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Biotech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 06-TLF-001
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-01

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OP-1 Putty (Experimental): Patients randomized to the OP-1 Putty Spinal System arm will receive OP-1 Putty with AVS™TL PEEK Spacer System and XIA® Spinal System.
  Interventions: Device: TLIF with a PEEK Spacer System and XIA Spinal System
- Autograft (Active Comparator): Patients randomized to the Autograft Spinal System arm will receive iliac crest autograft with AVS™TL PEEK Spacer System and XIA® Spinal System.
  Interventions: Device: TLIF with a PEEK Spacer System and XIA Spinal System

INTERVENTIONS:
Device: TLIF with a PEEK Spacer System and XIA Spinal System — TLIF with an AVS™TL PEEK Spacer System and XIA® Spinal System using either OP-1 Putty and/or Autograft.
  Other Names: TLIF with a Spacer System

SUMMARY:
This study will explore the use of recombinant OP-1 in conjunction with surgical treatment of single-level TLIF of the lumbar spine.

DETAILED DESCRIPTION:
This pilot study is a randomized, multi-center, prospective, controlled study of the efficacy and safety of OP-1 Putty Spinal System in patients requiring a single level transforaminal interbody fusion of the lumbar spine (TLIF).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing and able to understand, sign and date the study-specific, Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved patient informed consent and applicable privacy regulations.
2. The patient has a documented diagnosis of DDD with up to Grade I spondylolisthesis demonstrated by radiographic imaging (by plain film/discography within 12 weeks of surgery and/or computed tomography (CT scan/magnetic resonance imaging [MRI].
3. The patient requires single level lumbar fusion (L2 to S1)

Exclusion Criteria:

1. The patient has a history of previous surgery in the lumbar spine with or without attempted fusion {Note: a history of lumbar decompression surgery is permitted}.
2. The patient has Grade II, Grade III or Grade IV spondylolisthesis.
3. The patient has gross spinal instability measured on flexion/extension radiographs of >25% translation of the vertebrae, or ≥20 degrees of angular motion or has significant (>10%) scoliosis.
4. The patient is receiving treatment (before, during or after surgery) with a drug that interferes with bone metabolism or is being treated with a bone growth stimulator.
5. The patient has been treated in the last 6 months with radiation, chemotherapy, immunosuppression or systemic corticosteroids.
6. The patient has a history of, or has any malignancy or spinal tumor of any type, with the exception of a history of a treated basal or squamous cell carcinoma.
7. The patient is morbidly obese (defined as body mass index [BMI] > 35).
8. The patient currently uses tobacco products, within 3 weeks prior to time of treatment.
9. The patient is known to require at the time of treatment, additional surgery to the lumbar spinal region within the next 6 months or has symptomatic multilevel degenerative disease requiring possible instrumented fusion of more than one level.
10. The patient has previously been treated with or exposed to any Bone Morphogenetic Proteins (BMPs).
11. The patient is contraindicated for iliac crest autografting in that the Investigator believes the patient would be unable to provide sufficient quantity or adequate quality autograft (e.g., osteoporosis as defined by this protocol) from a unilateral iliac crest harvest.
12. The patient has a previous diagnosis of Paget's disease, osteomalacia or any other endocrine or metabolic bone disease that affects osteogenesis.
13. The patient has a documented history of osteoporosis or has a risk of osteoporosis as defined by an Osteoporosis Risk Assessment Instrument (ORAI) score of ≥ 9 and a DEXA Scan T score of ≥-2.5 standard deviations below the normal range within one year of enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pain and function as measured by an Oswestry Disability Index, no revisions, removals or supplemental fixations, fusion success, defined as radiographic evidence of fusion, maintenance or improvement in lower extremity neurologic function | 12 and 24 months post intervention

SECONDARY OUTCOMES:
Quality of life determinations (SF-36), pain assessments (VAS), work status and assessment of additional radiographic parameters | 12 and 24 months post intervention

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Los Angeles, California
  - San Diego, California
  - Durango, Colorado
  - Boston, Massachusetts
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Omaha, Nebraska
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Temple, Texas